CLINICAL TRIAL: NCT06492655
Title: A Randomized, Open-label, Single Dose, Crossover, Phase 1 Trial to Evaluate the Food Effect on Pharmacokinetic Profiles and Safety of CKD-383 in Healthy Volunteers
Brief Title: To Evaluate the Food Effect on Pharmacokinetic Profiles and Safety in Healthy Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A101_06FDI2404
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lobeglitazone; empagliflozin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Other): * Period 1: CKD-383 two tablets(Fed)
  * Period 2: CKD-383 two tablets(Fasted)
  Interventions: Drug: CKD-383(Fed); Drug: CKD-383(Fasted)
- Group 2 (Other): * Period 1: CKD-383 two tablets(Fasted)
  * Period 2: CKD-383 two tablets(Fed)
  Interventions: Drug: CKD-383(Fed); Drug: CKD-383(Fasted)

INTERVENTIONS:
Drug: CKD-383(Fed) — After maintaining NPO for at least 10 hours before a high-fat meal, take a high-fat meal within 20 minutes on each medication day, and take CKD-383 two tablets orally with 150 mL of water at room temperature.
  Other Names: Lobeglitazone, Empagliflozin, Metformin
Drug: CKD-383(Fasted) — After maintaining NPO for at least 10 hours before dosing, and take CKD-383 two tablets orally with 150 mL of room temperature water with 30g of sugar added on each dosing day.
  Other Names: Lobeglitazone, Empagliflozin, Metformin

SUMMARY:
This is a randomized, open-label, single dose, crossover, phase 1 trial to evaluate the food effect on pharmacokinetic profiles and safety of CKD-383 in healthy volunteers

DETAILED DESCRIPTION:
Participants were randomly assigned in a 1:1 ratio. TheParticipants are prescribed oral administration of the appropriate IP(2 tablets in single dose: actual medication)

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 19 to 54 years
* BMI measurement result is 18.0 kg/m2 to 30 kg/m2
* Written informed consent
* Other inclusion criteria, as defined in the protocol

Exclusion Criteria:

* who has taken drug metabolism enzyme induction and inhibitory drugs, such as barbitale drugs, within 30 days prior to the start of the trial (Period

  1 administration)
* Other exclusive criteria, as defined in the protocol

Ages: 19 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-07-04 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-08 (Estimated)

PRIMARY OUTCOMES:
AUCt of Empagliflozin, sitagliptin, metformin(Participants greater than or equal to 18.0 kg/m2 and less than 30 kg/m2) | 0 hour ~ 48 hour after drug administration
  Pharmacokinetic characterization
Cmax of Empagliflozin, sitagliptin, metformin(Participants greater than or equal to 18.0 kg/m2 and less than 30 kg/m2) | 0 hour ~ 48 hour after drug administration
  Pharmacokinetic characterization

CONTACTS AND LOCATIONS:
Overall Officials: Jaeyong chung, PI, Principal Investigator — Seoul National University Bundang Hospital

IPD SHARING:
Plan to Share IPD: No